CLINICAL TRIAL: NCT05491525
Title: A Phase 2/3, Open-label, Baseline-controlled, Multicenter, Long-term Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Vibegron in Pediatric Subjects 2 Years to < 18 Years of Age With Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)
Brief Title: A Study of Vibegron in Pediatric Participants 2 Years to Less Than (<) 18 Years of Age With NDO and on CIC
Acronym: KANGUROO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: URO-901-3007
Record Dates: First submitted 2022-07-28; First posted 2022-08-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Neurogenic Detrusor Overactivity; Vibegron; Clean Intermittent Catheterization; Beta-3 Adrenergic Receptor Agonist; Maximum Cystometric Capacity; Spinal Dysraphism; Spina Bifida; Myelomeningocele; Meningocele; Spinal cord injury; Transverse myelitis
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele; Meningocele; Spinal Cord Injuries; Myelitis, Transverse | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Vibegron Adolescents (12 to < 18 years) (Experimental): Part A: Participants aged 12 to < 18 years will receive vibegron based on their weight, with dose reduction based on individual clinical condition, PK, and safety/tolerability data. Participants may be dose-reduced up to 2 times.
  Part B: Participants will receive a Data and Safety Monitoring Board (DSMB)-selected vibegron dose for their weight determined from participants in their respective cohort and weight band of Part A.
  Interventions: Drug: Vibegron
- Cohort 2: Vibegron Children (2 to < 12 years) (Experimental): Part A: Participants aged 2 to < 12 years will receive vibegron based on their weight, after DSMB review of Cohort 1, Part A data, with dose reduction based on individual clinical condition, PK, and safety/tolerability data. Participants may be dose-reduced up to 2 times.
  Part B: Participants will receive a DSMB-selected vibegron dose for their weight determined from participants in their respective cohort and weight band of Part A.
  Interventions: Drug: Vibegron

INTERVENTIONS:
Drug: Vibegron — Participants will be administered Vibegron orally, once daily (QD)

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and PK of vibegron in pediatric participants with NDO who are regularly using CIC

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, age 2 years to < 18 years at the Screening Visit. Participants age 12 to < 18 years (Cohort 1) must weigh at least 29.5 kilograms (kg). Participants age 2 to < 12 years (Cohort 2) must weigh at least 11 kg.
* Participant has been diagnosed with NDO due to one of the following: spinal dysraphism, which includes spina bifida (eg, myelomeningocele, meningocele) and all forms of tethered cord; or acquired NDO from a spinal cord injury or spinal cord surgery, with the injury/surgery having occurred at least 6 months prior to the Screening Visit; or acquired NDO due to transverse myelitis with diagnosis at least 12 months prior to the Screening Visit.
* Participant undergoes CIC at least 3 times per 24 hours (with the last CIC performed prior to going to sleep for the night) for at least 4 weeks prior to the Screening Visit.

Exclusion Criteria:

* Participant has cerebral palsy, uncontrolled epilepsy, diabetes insipidus, or Stage 2 hypertension
* Participant has an active malignancy in the 12 months prior to the Screening Visit.
* Participant has been administered intravesical botulinum toxin within 9 months prior to the Screening Visit and should remain off this therapy during the study.
* Participant is taking digoxin or lithium within 10 days prior to Screening Visit or plans to start taking either during the study.
* Participant currently uses or plans to use a baclofen pump during the study.
* Participant has urethral dilatation or has had urethral surgery in the 3 months prior to the Screening Visit.
* Participant has undergone bladder augmentation surgery.
* Participant has a known genitourinary condition (other than NDO) that may cause overactive contractions or incontinence (bladder exstrophy, urinary tract obstruction, urethral diverticulum or fistula) or bladder stones or another persistent urinary tract pathology that may cause symptoms.
* Participant has an insufficient urethral sphincter, has had implantation of an artificial sphincter, has a surgically-treated underactive urethral sphincter, or, in the 6 months prior to the Screening Visit, has undergone pelvic gender reassignment surgery.
* Participant has one of the following gastrointestinal problems: partial or complete obstruction, decreased motility such as paralytic ileus, risk of gastric retention, or malabsorption syndrome of any form.
* Participant has fecal impaction or a history of fecal impaction requiring hospitalization or ambulatory surgical treatment in the 3 months prior to the Screening Visit.
* Participant has a urinary indwelling catheter in the 4 weeks prior to the Screening Visit.
* Participant has moderate to severe dilating vesicoureteral reflux (Grade III to V) or severe renal failure.
* Participant started electrostimulation/neuromodulation therapy in the 4 weeks before the Screening Visit, or is expected to start this therapy during the study period.
* Participant has participated in another clinical trial and/or has taken an investigational drug within 4 weeks prior to the Screening Visit.
* Participant is unable, or parent/caregiver is not willing, to washout any medication for the management of NDO.
* Participant is a female of childbearing potential who is unwilling or unable to use a highly effective method of contraception for the duration of the study.
* Female participants who are currently breastfeeding or plan to breastfeed any time from the Screening Visit until 28 days after the final study drug administration.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in maximum cystometric capacity (MCC) based on bladder filling urodynamics | Baseline and at Week 32

SECONDARY OUTCOMES:
Change from Baseline in MCC | Baseline and at Week 20
Change from Baseline in number of overactive detrusor contractions until the end of bladder filling | Baseline and at Weeks 20 and 32
Change from Baseline in detrusor pressure at the end of bladder filling | Baseline and at Weeks 20 and 32
Change from Baseline in bladder filling volume until first involuntary/hyperactive detrusor contraction | Baseline and at Weeks 20 and 32
Change from Baseline in bladder compliance (mL/cm H2O) | Baseline and at Weeks 20 and 32
  Bladder compliance is calculated by dividing the change in volume by the change in detrusor pressure during the filling of the bladder
Change from Baseline in average first morning catheterized volume | Baseline and at Weeks 1, 4, 8, 20, 32, 48, and 52
Change from Baseline in average catheterized volume per catheterization | Baseline and at Weeks 1, 4, 8, 20, 32, 48, and 52
Change from Baseline in average maximum catheterized volume per day | Baseline and at Weeks 1, 4, 8, 20, 32, 48, and 52
Change from Baseline in average maximum catheterized daytime volume | Baseline and at Weeks 1, 4, 8, 20, 32, 48, and 52
Change from Baseline in average number of leakage episodes per day | Baseline and at Weeks 1, 4, 8, 20, 32, 48, and 52
Change from Baseline in estimated number of dry (leakage-free) days/ 7 days | Baseline and at Weeks 1, 4, 8, 20, 32, 48, and 52
Change from Baseline in Pediatric Incontinence Questionnaire (PIN-Q) | Baseline and at Weeks 20, 32 and 52
  PIN-Q is a 20-item questionnaire addressing quality of life for participants with bladder disorders. Each question was answered on a scale from 0 (no, never) to 4 (all the time). The total score ranged from 0 to 80, with higher scores indicating more impact on the quality of life.
Change from Baseline in Patient Global Impression of Severity (PGI-S) Scale | Baseline and at Weeks 20, 32 and 52
  PGI-S is a 5 point scale that determines the bladder condition of a participant with 0 being really bad and 4 as really good. Higher score indicates better bladder condition.
Change from Baseline in Clinical Global Impression of Change (CGI-C) Scale | Baseline and at Weeks 20, 32 and 52
  The CGI-C scale is used to determine the degree of change in participant's overall bladder symptoms since the start of the study on Day 1. The scale will be filled by the investigator by ticking on any of the following options: very much improved, much improved, minimally improved, no change, minimally worse, much worse and very much worse.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Children's Hospital of Orange County, Orange, California
  - Nemours Childrens Health, Jacksonville, Jacksonville, Florida
  - Wichita Urology Group, Wichita, Kansas
  - Childrens Hospital New Orleans, New Orleans, Louisiana
  - Albany Medical College, Albany, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Urovant is committed to sharing patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Data requests will be reviewed and approved on the basis of scientific merit. All data provided will be anonymized according to applicable laws and regulations.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be made available within 24 months after study completion and will be accessible for a time frame appropriate for the approved proposal.
Access Criteria: Access to these clinical trial data can be requested by emailing medinfo@urovant.com and will be provided following Urovant review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).